CLINICAL TRIAL: NCT04132076
Title: Treatment Outcome After Ankle Joint Surgeries
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Urban Brulc, Medical doctor, resident of orthopaedic surgery, University Medical Centre Ljubljana
Other Study IDs: 0120-99/2019/4
Record Dates: First submitted 2019-10-13; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Osteochondral Lesion of Talus; Ankle Arthritis; Instability; Ankle (Ligaments) (Old Injury); Impingement Syndrome of Ankle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Osteochondral lesion of talus (OLT): Patients with OLT treated operatively (debridement, microfracture, allograft, mesenchymal stem cells implantation) in Department of Orthopaedic Surgery, University Medical Centre Ljubljana (UMC).
- Group B: Ankle joint osteoarthrosis: Patients with ankle joint osteoarthrosis treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.
- Group C: Ankle Impingement syndrome: Patients with ankle impingement syndrome treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.
- Group D: Ankle instability syndrome: Patients with ankle instability syndrome treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.

SUMMARY:
Osteochondral lesion of talus (OLT), osteoarthrosis and impingement/instability syndrome are most common ankle joint pathologies. This study analyses outcome after various different operative treatment of aforementioned pathologies. Investigators hypothesis is that patient characteristics, type of lesion and surgical technique affect the result of treatment. The investigators will compare subjective (questionnaire) and objective (clinical examination) status of patient before and after operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OLT treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.
* Patients with ankle joint osteoarthritis treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.
* Patients with ankle instability syndrome treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.
* Patients with ankle impingement syndrome treated operatively in Department of Orthopaedic Surgery, UMC Ljubljana.

Exclusion Criteria:

* patient refuse to participate in study
* no respond of patient after invitation to answer a standardized questionnaire (EQ-5D, FAOS, Tegner activity score)
* no respond of patient after invitation to control examination after operation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The invetigators will analyse cohort of patient after ankle joint surgery in the Department of Orthopaedic Surgery, UMC Ljubljana between 2008 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
FAOS questionnaire | 36 months after operation
  Foot and Ankle Outcome Score (FAOS) is a patient reported instrument that may be useful for assessing changes in foot/ankle pathology over time, with or without treatment. It assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and foot/ankle related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible foot/ankle symptoms and 100 indicating no foot/ankle symptoms.
EQ-5D questionnaire | 36 months after operation
  EQ-5D is a standardized instrument for measuring generic health status. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale used in the health state description part has three-level; having no problems, having some or moderate problems, being unable to do/having extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).
Tegner activity score | 36 months after operation
  Tegner activity score is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity. The score varies from 0-10. A score of 0 represents sick leave or disability pension, whereas a score of 10 corresponds to participation in national and international elite competitive sports.

SECONDARY OUTCOMES:
Kellgren and Lawrence score | 36 months after operation
  Kellgren and Lawrence score is a common method of classifying the severity of osteoarthritis (OA) using five grades.
  grade 0: no radiographic features of OA are present grade 1: doubtful joint space narrowing (JSN) and possible osteophytic lipping grade 2: definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph grade 3: multiple osteophytes, definite JSN, sclerosis, possible bony deformity grade 4: large osteophytes, marked JSN, severe sclerosis and definite bony deformity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of orthopaedic surgery, University medical centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Kolar M, Brulc U, Strazar K, Drobnic M. Patient-reported joint status and quality of life in sports-related ankle disorders and osteoarthritis. Int Orthop. 2021 Apr;45(4):1049-1055. doi: 10.1007/s00264-020-04747-y. Epub 2020 Sep 17. PMID 32944803